

# CLINICAL STUDY PROTOCOL: OTL-2016-OTL38-005

| Title: | A Phase 2, Single dose, Open-Label, Exploratory Study to<br>Investigate the Safety and Efficacy of OTL38 Injection for<br>Intraoperative Imaging of Folate Receptor Positive Lung Nodules |
|---|---|
| Test Drug: | OTL38 Injection: folate analog ligand conjugated with an indole cyanine-like green dye as a solution in vials containing 1.6 mL at 2 mg/mL |
| Protocol Identification: | OTL-2016-OTL38-005 |
| Sponsor Name and Address: | On Target Laboratories, Inc. |
| Compliance Statement: | The study will be conducted in accordance with standards of Good Clinical Practice, as defined by the International Conference on Harmonisation and all applicable national and local regulations. |
| Date of Protocol<br>Amendment: | Version 5.0, 14 June 2018 |
| | Signature |

## CONFIDENTIALITY STATEMENT

The information contained within this report is confidential and may not be used, divulged, published, or otherwise disclosed without the prior written consent of On Target Laboratories, Inc.

#### **Medical Monitor Contact:**

| Name: | |
|----------|----|
| Address: | 27 |
| Phone: | |
| Fax: | |
| E-mail: | |

## **Sponsor Contact:**

| Name: |
|----------|
| Address: |
| Phone: |
| Fax: |
| E-mail: |

## **Sponsor Regulatory Contact:**

| Name: |
|----------|
| Address: |
| Phone: |
| Fax: |
| E-mail: |

Medelis, Inc. will notify the On Target US Regulatory representative, any SAE/SUSAR/unanticipated ADE report that it receives. In addition, will provide to On Target Regulatory the initial documents regarding a SAE/SUSAR/unanticipated ADE and follow-up documents regarding each event on proper FDA forms. This information will be supplied to On Target expeditiously in order for On Target to submit the safety information to the FDA within the safety reporting time regulations.

will notify all sites of any SAE/SUSAR/unanticipated ADE report it receives. It is each Investigator's responsibility to forward to the site's IRB/EC all SAE/SUSAR/unanticipated ADE reports from other sites that are transmitted on behalf of the Sponsor by


# SERIOUS ADVERSE EVENT, SUSPECTED UNEXPECTED SERIOUS ADVERSE REACTIONS, AND UNANTICIPATED ADVERSE DEVICE EFFECT REPORTING

| CONTACT | WITHIN 24 HOURS OF LEARNING OF ANY SERIOUS |
|---|---|
| | SERIOUS ADVERSE REACTIONS AND UNANTICIPATED |
| | <u>DVERSE</u> EVENT IS FATAL OR LIFE THREATENING, THE |
| SPONSOR AND | MUST BE INFORMED IMMEDIATELY. |
| Complete and fax a Serious Adverse | Event report form and provide any supporting |
| documentation to | as described below: |
| | do 333113 3 3 3 3 1 1 1 1 1 1 1 1 1 1 1 1 |
| | A |
| SAFETY SURVEILLANCE: | MEDICAL MONITOR |
| SAFETT SURVEILLANCE. | MEDICAL MONTOR |
| | • |

To discuss SAE with the Medical Monitor, contact at the numbers provided above.

Follow-up information to serious AEs must be provided to within 24 hours of investigator awareness in the same manner detailed above.


# 1 PROTOCOL SYNOPSIS

| Study Title | A Phase 2, Single dose, Open-Label, Exploratory Study to Investigate the Safety and Efficacy of OTL38 Injection for Intraoperative Imaging of Folate Receptor Positive Lung Nodules |
|---|---|
| Protocol Number | OTL-2016-OTL38-005 |
| Sponsor | On Target Labs, Inc. |
| Investigational<br>Product | OTL38 Injection: folate analog ligand conjugated with an indole cyanine-like green dye as a solution in vials containing 1.6 mL at 2 mg/mL |
| Primary<br>Objectives | <ul> <li>To estimate the Sensitivity and False Positive rate of OTL38 for malignancy detection during Near Infrared Imaging (NIR).</li> <li>To assess the safety and tolerability of single intravenous doses of OTL38.</li> </ul> |
| Secondary<br>Objectives | <ul> <li>To assess the safety of the Fluorescence Imaging Systems for intraoperative imaging when used with OTL38.</li> <li>To estimate the efficacy of OTL38 and NIR with respect to the identification of Clinically Significant Events (CSEs).</li> </ul> |
| Exploratory | |
| Study Design | This is a phase 2, multi-center, single dose, open-label, exploratory study in suspected lung cancer patients scheduled to undergo endoscopic or thoracic surgery per CT/PET imaging based on standard of care. |
| Treatment | <ul> <li>OTL38 is a folate analog ligand conjugated with an indole cyanine-like green dye.</li> <li>Each patient will be administered a single dose of OTL38 and study-related procedures will last from approximately 2-3 hours before dosing to 24 hours after dosing.</li> <li>The imaging systems used in this study are not approved for use with OTL38, and are therefore considered investigational for the purposes of this study (see Section 5.8.5 for additional information) Full specifications for</li> <li>The imaging system used by the investigational site will be recorded in the eCRF.</li> </ul> |


| Study Duration | • Patients will complete a single dose of OTL38 initiation of intraoperative imaging. |
|---|---|
| | • Safety assessments: during infusion of OTL38; post-surgery; Day 7 (± 4), and Day 28 (± 7) after surgery. |
| | • Estimated total length of study: 18 months |
| | • Patient accrual estimate: 12 months |
| Eligibility | Inclusion: |
| Criteria | 1. Male and Female patients 18 years of age and older |
| | 2. Confirmed diagnosis of adenocarcinoma lung cancer |
| | OR, |
| | 3. Have a primary diagnosis, or at high clinical suspicion, of lung nodule(s) warranting surgery based on CT and/or PET imaging |
| | 4. Who are scheduled to undergo endoscopic or thoracic surgery |
| | 5. A negative serum pregnancy test at Screening followed by a negative urine pregnancy test on the day of surgery or day of admission for female patients of childbearing potential |
| | 6. Female patients of childbearing potential or less than 2 years postmenopausal agree to use an acceptable form of contraception from the time of signing informed consent until 30 days after study completion |
| | 7. Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and to return for the required assessments |
| | Exclusion: |
| | 1. Previous exposure to OTL38 |
| | 2. Known FR-negative lung nodules |
| | 3. Any medical condition that in the opinion of the investigators could potentially jeopardize the safety of the patient |
| | 4. History of anaphylactic reactions |
| | 5. History of allergy to any of the components of OTL38, including folic acid |
| | 6. Pregnancy, or positive pregnancy test |
| | 7. Clinically significant abnormalities on electrocardiogram (ECG) at screening. |
| | 8. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule |
| | 9. Impaired renal function defined as eGFR< 50 mL/min/1.73m2 |
| | 10. Impaired liver function defined as values > 3x the upper limit of normal (ULN) for alanine aminotransferase (ALT) or aspartate aminotransferase (AST), alkaline phosphatase (ALP), or total bilirubin. |
| | 11. Received an investigational agent in another investigational drug or vaccine trial within 30 days prior to surgery |
| | 12. Known sensitivity to fluorescent light |
| Number of<br>Subjects | Up to 110 patients with suspected lung cancer will be enrolled in this study |


| Number of | Up to six (6) investigational sites: |
|---|---|
| Investigator Sites | University of Pennsylvania University of Pittsburgh Medical Center |
| | Beth Israel Deaconess Medical Center |
| | MD Anderson Cancer Center |
| | Leiden University Medical Center Cleveland Clinic |
| 7 M 8 1929 | . 7 1 2 2 2 1 1 1 1 2 2 2 2 2 2 2 2 2 2 2 |
| Assessments | Visit 1-Screening (up to 28 days prior to surgery): |
| | Signed informed consent |
| | Complete medical history |
| | Physical examination |
| | Height and weight |
| | Concomitant medication assessment |
| | Vital signs (temperature, blood pressure, and pulse rate) |
| | Serum Pregnancy test (for women of childbearing potential) |
| | • 12-lead ECG |
| Clinical laboratory assessments including hematology, chemistries, ar analysis | |
| | Visit 2-Day of Admission (Day 0) or Day of Surgery (Day 1): |
| | Updated medical history and physical exam |
| | Concomitant medications assessment |
| | Clinical Laboratory and vital sign assessments will be performed |
| | • Urine pregnancy test (for women of childbearing potential) |
| | • 12- Lead ECG will be collected at least 15 minutes prior to infusion, and at least 15 minutes prior to surgery after infusion of OTL38 is completed |
| | A single dose of OTL38 will be infused IV over approximately 60 minutes initiation of intraoperative imaging and the time will be recorded |
| | AEs will be recorded during infusion of OTL38 |
| | During and post-surgery any AEs and ADEs will be recorded. |
| | Day 1 - Surgery |
| | At least one hour prior to initiation of intraoperative imaging, patients will complete an infusion of of OTL38. |














## Visit 3-Follow-up (Day 7 [ $\pm$ 4]):

- Follow-up will be scheduled for Day 7 ( $\pm$  4) on site
- AEs, ADEs, and concomitant medication information will be recorded.
- Clinical laboratory and vital sign assessments will be performed.

## Visits 4-Follow-up (Day 28 $[\pm 4]$ ):

- Follow-up will be scheduled for Day 28 (±4) either via patient telephone interview or clinic visit
- AEs, ADEs, and concomitant medication information will be collected.

#### **Study Endpoints**

#### Primary

The primary efficacy endpoints are the Sensitivity and False Positive rate of OTL38 for malignancy detection during Near Infrared Imaging (NIR).



### Secondary

The secondary efficacy endpoint is proportion of patients with at least one CSE as a result of utilizing OTL-38 and Near Infrared Imaging.







| Statistical<br>Methods | Primary Efficacy Endpoints Given the design of the study the primary focus of the analysis will be estimation rather than hypothesis testing. |
|---|---|
| Safety | Safety will be described via subject incidence of treatment emergent adverse events (TEAEs) including serious TEAEs as well as adverse device effects (ADEs). Additionally, summary statistics and/or shift tables will be provided for vital signs, physical exams, ECGs, and laboratory parameters at baseline and post-baseline measurements. |
| | Further analytic details for efficacy and safety will be provided in the statistical analysis plan (SAP). |


# 2 SCHEDULE OF PROCEDURES


# **Table of Contents**

| 1 | PRO | OTOCOL SYNOPSIS | 4 |
|---|---|---|---|
| 2 | SCH | HEDULE OF PROCEDURES | 14 |
| 3 | BAC | CKGROUND INFORMATION | 19 |
| | 3.1 | Background | 19 |
| | 3.2 | Rationale | 19 |
| | 3.3 | Investigational Product | 20 |
| | | 3.3.1 Prior Clinical Experience | |
| | | 3.3.2 Phase 1b Ovarian Cancer Study (CHDR1321-B) | |
| | | 3.3.3 Phase 2 Ovarian Cancer Study (OTL-2016-OTL38-0 | 03)21 |
| | | 3.3.4 Early Clinical Experience with Lung and Pituitary pa | atients:21 |
| | 3.4 | Risks and Benefits of OTL38 | 22 |
| | | 3.4.1 Risks | 22 |
| | | 3.4.2 Benefits | 23 |
| 4 | STUDY OBJECTIVES24 | | |
| | 4.1 | Primary | 24 |
| | 4.2 | • | |
| | 4.3 | Exploratory | |
| 5 | STU | STUDY DESIGN | |
| | 5.1 | Overall Investigation Plan | |
| | | 5.1.1 Safety assessment | |
| | | 5.1.2 Tumor to Background Ratio | |
| | 5.2 | Eligibility Criteria | |
| | 0.2 | 5.2.1 Inclusion Criteria | |
| | | 5.2.2 Exclusion Criteria | |
| | 5.3 | Study Assessments | |
| | 5.4 | <del>-</del> | |
| | 5.5 | | |
| | 5.6 | | |
| | 2.0 | 5.6.1 Identification and Description of Test Article | |
| | | 5.6.2 Packaging and Labeling | |
| | | 5.6.3 Storage and Handling of Test Article | |
| | | 5.6.4 Study Drug Administration | |
| | | 5.6.5 Camera/Imaging System | |

| | | | 5.6.5.1 Summary of the Camera/Imaging System Requirem | ents29 |
|---|---|---|---|---|
| | | | 5.6.5.2 Quality System Requirements | 30 |
| | 5.7 | Conco | omitant Medications | 31 |
| | | 5.7.1 | Allowed Medications | 31 |
| | | 5.7.2 | Prohibited Medications | 31 |
| | 5.8 | Sched | ule of Events | 31 |
| | | 5.8.1 | Measurement and Evaluations | 31 |
| | | | 5.8.1.1 Visit 1 (Screening, up to Day -28) | 31 |
| | | | 5.8.1.2 Visit 2- Day of Surgery (Day 1): | 32 |
| | | | 5.8.1.3 Visit 3-Follow-up (Day 7 [± 4]): | 36 |
| | | | 5.8.1.4 Visits 4-Follow-up (Day 28 [±4]): | |
| | | 5.8.2 | Surgical Reporting Schematic | |
| | | 5.8.3 | Post-Surgery Questionnaire | |
| | | 5.8.4 | Pathology Samples | |
| | | 5.8.5 | Camera/Imaging System Exposure | |
| 6 | STU | STUDY ENDPOINTS | | |
| | 6.1 | Effica | cy | 38 |
| | 6.2 | Second | dary Efficacy | 38 |
| | 6.3 | Explo | ratory | 39 |
| | 6.4 | Safety | <i>T</i> | 39 |
| 7 | PROCEDURES FOR REPORTING ADVERSE EVENTS | | | |
| | 7.1 | Adverse Events Definitions | | |
| | 7.2 | 7.2 Adverse Device Effects Definitions | | |
| | | 7.2.1 | Adverse Device Effect | 40 |
| | | | 7.2.1.1 Suspected Adverse Device Effect | 41 |
| | | | 7.2.1.2 Unanticipated Adverse Device Effect | 41 |
| | 7.3 | Report | ting of Adverse Events | 41 |
| | | 7.3.1 | Adverse Events | 41 |
| | | 7.3.2 | Laboratory Abnormalities | 41 |
| | | 7.3.3 | Serious Adverse Events | 42 |
| | | 7.3.4 | Reporting of Pregnancies | 42 |
| | | 7.3.5 | Disease Progression | 42 |
| | | 1.1.1 | Overdoses | 42 |
| | 7.4 | Classi | fication of Adverse Events by Severity | 42 |
| | 7.5 | Classi | fication of Adverse Events by Relationship to Study Drug Admir | nistration43 |
| | 7.6 | Advers | rse Events Qualifying for Expedited Reporting | 43 |

| 8 | DAT | A REC | <b>ORDING</b> | , CRF PROCESSING, AND STATISTICAL ANALYSIS | 44 |
|---|---|---|---|---|---|
| | 8.1 Data Recording and CRF Processing | | | | 44 |
| | 8.2 | Statistical Methods | | | |
| | | 8.2.1 Sample Size Estimation | | | |
| | | 8.2.2 | Analysis Sets Description of Subgroups to be Analyzed | | 45 |
| | | 8.2.3 | | | 45 |
| | | 8.2.4 | | | 46 |
| | | 8.2.5 | Statistical Analysis | | |
| | | | 8.2.5.1 | Primary Efficacy Endpoints | 46 |
| | | | 8.2.5.2 | Secondary Efficacy Endpoint | |
| | | | 8.2.5.3 | Safety Evaluations | 47 |
| | | | 8.2.5.4 | Imaging System | 48 |
| | | | 8.2.5.5 | Prior and Concomitant Medications | |
| | | | 8.2.5.6 | Handling of Missing Data, Subject Withdrawals, and Treatr Failures | |
| | | | 8.2.5.7 | Interim Analyses | 49 |
| 9 | ETH | ICS | •••• | | 50 |
| | 9.1 | Patient | Informati | ion and Consent | 50 |
| | 9.2 | Institutional Review Board | | | |
| 10 | STUDY ADMINISTRATION | | | | |
| | 10.1 | | | | |
| | 10.2 | Study Record Retention | | | |
| | 10.3 | Patient | ity | 51 | |
| | 10.4 | | | | |
| 11 | INVI | ESTIGA | ATOR'S S | STATEMENT | 52 |
| 12 | | | | | |
| AII | | ICES | ••••• | | JT |
| | | | | Table of Figures | |
| T2: - | 1 | TDI | ) I | _ | 25 |
| _ | ire 1. | | | 1E : G . COTI 10 | |
| Figure 2. | | | Excitation and Emission Spectra of OTL38 | | |
| Figure 3. | | Clas | ssification | Table | 46 |


# **List of Abbreviations**

| Abbreviation | Definition |
|---|---|
| ADE | Adverse Device Effect |
| AE | Adverse Event |
| AEL | Accessible Emission Limits |
| ALT (SGPT) | Alanine aminotransferase (serum glutamic pyruvate transaminase) |
| AST (SGOT) | Aspartate aminotransferase (serum glutamic oxaloacetic transaminase) |
| BUN | Blood urea nitrogen |
| CFR | Code of Federal Regulations |
| CSE | Clinically Significant Event |
| EC | Ethics Committee |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| FDA | United States Food and Drug Administration |
| FITC | Fluorescein isothiocyanate |
| FN | False Negative |
| FP | False Positive |
| FR | Folate Receptor |
| GCP | Good Clinical Practice |
| IB | Investigator Brochure |
| ICH | International Conference on Harmonisation |
| IND | Investigational New Drug |
| IRB | Institutional Review Board |
| MedDRA | Medical Dictionary for Regulatory Activities |
| SAE | Serious adverse event |
| SUSAR | Suspected unexpected serious adverse reaction |
| TAM | Tumor Associated Macrophages |
| TEAE | Treatment Emergent Adverse Event |
| TN | True Negative |
| TP | True Positive |
| ULN | Upper limit of the normal range |
| WHO | World Health Organization |


## 3 BACKGROUND INFORMATION

# 3.1 Background

According to the World Health Organization, lung cancer is the leading cause of cancer-related deaths in men and women, and is responsible for 1.6 million deaths worldwide annually as of 2012 (Stewart 2014). Surgery remains the preferred method of treatment and the only potentially curative modality for patients presenting with operable Stage I or II lung cancers; however, the 5-year survival rates for these candidates remain at 55.2% and 28.0% for Stages I and II lung cancer, respectively (SEER 2016). These high rates of local recurrence may be due to the inability to completely detect and remove primary tumor nodules, and lingering metastases in synchronous nodules (tumors located within proximal parenchyma) in a satisfactory manner. Eliminating positive tumor margins through imaging during surgery could facilitate improved rates of recurrent-free patients and thus overall survival (Okusanya 2014, Keating 2015).

## 3.2 Rationale

Approximately 85% of lung and pleural malignancies express folate receptor positive nodules (FR+), thus making folate receptors (FR) ideal targets for imaging agents such as OTL-38 (Shen 2015). OTL38 has been observed in preliminary Investigator Initiated studies as being effective in identifying non-malignant lung nodules. These nodules (such as granulomas) do not necessarily pose a threat to the patient's life, but are still targeted for removal by a surgeon to confirm the absence of cancer. Both malignant adenocarcinoma and benign lung nodules that fluoresce in situ are noted to have infiltrates of tumor associated macrophages (TAMs) expressing FR on immunohistochemistry (Shen 2015, De Jesus 2015). Therefore, this intraoperative imaging of lung cancers and nodules would be well-suited in the reduction of positive margins, identification of synchronous lesions, localization of sub-centimeter nodule and tumor tissue, and potentially improving clinical outcomes in these patients. Chemotherapy does not appear to affect FR expression in cancer specimens as examined by immunohistochemistry thus prior treatment is unlikely to affect utility of FR ligands as imaging agents (Crane 2012, Okusanya 2014). Since FRα is normally expressed only in the proximal tubules of the kidneys and in the choroidal plexus, uptake of OTL-0038 in the kidneys is possible (Ross 1994). However, the imaging described in this protocol will not involve tissue proximal to the kidneys.

While folate will initially distribute to all cells, redistribution, metabolism, and excretion will eliminate most of this agent from healthy tissues within 2-3 hours. Tumor cells that over expresses FR will retain folate and any fluorescent labeled folate conjugate (Leamon 1993). On Target Laboratories, Inc. has developed OTL0038, a folate analog ligand conjugated with an indole cyanine-like green dye developed by On Target Laboratories, Inc. as a tumor-imaging agent for patients with tumors that overexpress FRα.


## 3.3 Investigational Product

The resulting imaging agent, OTL0038 (also known as OTL-0038 or OTL-038), is the active pharmaceutical ingredient (API) of the drug product, OTL38 Injection (also known as OTL38). All nonclinical studies were conducted with API (drug substance) while clinical studies used OTL38 Injection.



The safety profile of OTL0038 has been characterized in a comprehensive series of non-human pharmacokinetic and toxicology studies. The results of the OTL0038 Phase 1-enabling nonclinical safety program in rats and dogs demonstrated the safe use of OTL0038 as an intraoperative imaging agent.

## 3.3.1 Prior Clinical Experience

OTL has completed a Phase 1A clinical trial to assess the safety, tolerability and pharmacokinetics of a single IV dose of OTL38 in healthy patients, a Phase 1b study of OTL38 for intraoperative imaging of FR $\alpha$  positive ovarian cancer, and a Phase 2 trial to investigate the safety and efficacy of OTL38 Injection for intraoperative imaging of FR $\alpha$  positive ovarian cancer.



# 3.3.2 Phase 1b Ovarian Cancer Study

Ten patients reported a total of 35 adverse events. The most common adverse events were post-surgical wound pain/discomfort, fatigue, abdominal pain/discomfort, nausea and vomiting. All events were graded as mild and all resolved within 1 day of the administration of OTL38. The majority of events were assessed as unrelated by the investigator and only two events (nausea and vomiting in the same) required action to be taken (administration of ondansetron).

No deaths occurred during the study. One patient who received a dose of developed two serious adverse events consisting of post-operative hospital-acquired pneumonia requiring antibiotics and coughing-induced wound dehiscence requiring surgical repair. These events were considered unrelated to OTL38 administration.




3.3.4 Early Clinical Experience with Lung and Pituitary patients:






Please refer to the Investigator's Brochure for more detailed information on OTL0038 and OTL38 Injection.

### 3.4 Risks and Benefits of OTL38

#### 3.4.1 Risks

The issues of possible concerns with the use of the OTL38 imaging systems are:

- Presence of an imaging system in the operating room
- Phototoxicity or thermal damage from the light source
- Nonspecific localization of OTL38
- Failure of OTL38 to bind to receptors
- Fading of the chromophore (photobleaching)
- Inability to excite the dye in OTL38 or to record emission
- Adverse events suggestive of hypersensitivity






#### 3.4.2 Benefits

The potential benefits of OTL38 for lung nodule imaging are:

- Improved staging of the tumor.
- Removal of additional lesions not previously noted on CT/PET
- Added assurance of clean margins to excised tumors.

In a preliminary investigator initiated study of OTL38 by Singhal et.al (2016 Pending), 8/47 (17.4%) of patients demonstrated a clinically significant event (CSE). A CSE is an occurrence that **would** result in modifying the scope or scale of an operation. By reducing the scale of an operation, patient morbidity could be decreased and recovery times improved. If other nodules are found in the chest cavity by NIR and are resected, this could prevent a recurrence of said cancer and significantly improve 5-year survivability. Further, recurrence prevention could preclude a patient from having to return to the hospital to have a second surgery scheduled.

This would need to be studied with other centers and physicians and in a larger patient population. Use of OTL38 would not change the surgeon's option to remove additional tissue because of impressions based on experience, visualization, or tactile senses.


## 4 STUDY OBJECTIVES

# 4.1 Primary

- To estimate the Sensitivity and False Positive rate of OTL38 for malignancy detection during Near Infrared Imaging (NIR).
- To assess the safety and tolerability of single intravenous doses of OTL38

## 4.2 Secondary

- To assess the safety of the Fluorescence Imaging Systems for intraoperative imaging when used with OTL38.
- To estimate the efficacy of OTL38 and Near Infrared Imaging (NIR) with respect to the identification of Clinically Significant Events (CSEs)

# 4.3 Exploratory




## 5 STUDY DESIGN

## 5.1 Overall Investigation Plan

This is a phase 2, multi-center, single dose, open-label, exploratory study in patients with folate receptor positive lung nodules scheduled to undergo endoscopic or thoracic surgery per CT/PET imaging based on standard of care. This includes wedge resection, lobectomy and thoracotomy and/or completion pneumonectomy.



## 5.1.1 Safety assessment

At each site, investigators will image their first patient meeting inclusion and exclusion criteria under the guidance of a surgeon trained in the use of the imaging agent and NIR camera system. The purpose of this training is to ensure correct use and operation of the camera system.

## 5.1.2 Tumor to Background Ratio

For cameras that are capable of doing so, tumor-to-background ratio will be calculated for each patient for comparison


## 5.2 Eligibility Criteria

## 5.2.1 Inclusion Criteria

To be considered eligible to participate in this study, a patient must meet all the inclusion criteria listed below:

- 1. Male and Female patients 18 years of age and older
- 2. Confirmed diagnosis of adenocarcinoma of the lung,

OR,

- 3. Have a primary diagnosis/high clinical suspicion of lung nodule(s) warranting surgery based on CT and/or PET imaging.
- 4. Scheduled to undergo endoscopic or thoracic surgery
- 5. A negative serum pregnancy test at Screening followed by a negative urine pregnancy test on the day of surgery or day of admission for female patients of childbearing potential
- 6. Female patients of childbearing potential or less than 2 years postmenopausal agree to use an acceptable form of contraception from the time of signing informed consent until 30 days after study completion
- 7. Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and to return for the required assessments

#### **5.2.2** Exclusion Criteria

Patients will be excluded if they meet any of the exclusion criteria listed below:

- 1. Previous exposure to OTL38
- 2. Known FR-negative lung nodules.
- 3. Any medical condition that in the opinion of the investigators could potentially jeopardize the safety of the patient
- 4. History of anaphylactic reactions
- 5. History of allergy to any of the components of OTL38, including folic acid
- 6. Pregnancy, or positive pregnancy test
- 7. Clinically significant abnormalities on electrocardiogram (ECG) at screening.
- 8. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
- 9. Impaired renal function defined as eGFR< 50 mL/min/1.73m<sup>2</sup>


- 10. Impaired liver function defined as values > 3x the upper limit of normal (ULN) for alanine aminotransferase (ALT) or aspartate aminotransferase (AST), alkaline phosphatase (ALP), or total bilirubin.
- 11. Received an investigational agent in another investigational drug or vaccine trial within 30 days prior to surgery.
- 12. Known sensitivity to fluorescent light

## 5.3 Study Assessments

The assessments for this study are listed in Section 5.8.

### 5.4 Patient Discontinuation Criteria

Although a single dose of study drug is infused on Day 1, a patient may be withdrawn from the study for any of the following reasons:

- Request of the patient or patient's representative
- AEs or adverse device effects (ADEs) based on the judgment of the Investigator
- The Investigator decides that it is in the patient's best interest
- The patient is noncompliant with the protocol
- Lost to follow-up
- Death

If a subject is withdrawn at any time, the reason(s) will be recorded on the relevant page of the electronic case report form (eCRF).

Patients discontinued due to AEs or ADEs will be monitored until resolution or stability of the event based on the judgment of the investigator.

# 5.5 Replacement of Dropouts

Patients withdrawing for reasons other than AEs or any other tolerability issues with the treatment may be replaced.

# 5.6 Study Drug Information and Dosage

# **5.6.1** Identification and Description of Test Article

OTL38 will be supplied in vials containing 1.6 mL of solution of 2 mg/mL OTL38 for a total of 3.2 mg of drug per vial.

Study medication should be stored in a freezer light (see Site Study Reference Manual).


A Research Pharmacist or other trained and qualified healthcare professional will prepare the IV solutions according to instructions provided by On Target Laboratories at the assigned dose. All prepared solutions should be protected from light (see Site Study Reference Manual) and refrigerated (between 2-8°C) until use.

## 5.6.2 Packaging and Labeling

The study medication will be packaged in vials and labelled by the Sponsor's clinical supplies designee.

The labels will include:

Name and contact information for the Sponsor:

Route of administration: injection

Quantity supplied: 3.2 mg OTL38 per vial

Pharmaceutical dosage form:

Storage conditions: keep frozen at temperature

CAUTION: New Drug - Limited by Federal Law To Investigational Use

Lot number

Manufacturing date in day/month/year format.

# 5.6.3 Storage and Handling of Test Article

The study medication will be packaged in vials and labelled by the Sponsor's clinical supplies designee.

## 5.6.4 Study Drug Administration

OTL38 will be prepared following the Dose Preparation for OTL38 Injection Pharmacy Manual (see Appendix 1). OTL38 will be administered intravenously over approximately 60 minutes, the infusion will be completed at least initiation of intraoperative imaging.

Intraoperative imaging beginning infusion will be considered a protocol deviation.







# 5.6.5.2 Quality System Requirements

On Target Laboratories outsources design and contract manufacturing for the final device and its labeling, and packaging. As part of the On Target Laboratories Supplier Approval Process, the contract manufacturer's quality system and compliance with the following federal and international regulations are assessed:

 USA 21 CFR Part 820: Code of Federal Regulations, Quality System Regulations; current edition


- ISO 13485:2003 Medical Devices Quality management systems Requirements for regulatory purposes
- Medical Device Directive: Council Directive 93/42/EEC concerning medical devices

### 5.7 Concomitant Medications

#### 5.7.1 Allowed Medications

Necessary supportive measures for optimal medical care will be given throughout the study. Additional care may be administered as indicated by the treating physician and patient's medical need, and after discussion with the medical monitor.

All concomitant medications and supportive therapy administered starting Day 1 prior to the infusion of OTL38 until the final study visit must be recorded on the appropriate case report form (eCRF).

#### 5.7.2 Prohibited Medications

No other investigational products will be allowed during this study. If the patient is on any folate supplement (including multi-vitamin supplements or pre-natal vitamins), the patient will need to stop taking the supplement 48 hours before scheduled drug infusion/surgery.



#### 5.8 Schedule of Events

#### 5.8.1 Measurement and Evaluations

Please see "Schedule of Events" for a detailed study schedule, including all measurements and evaluations for the entire study period (Screening to Follow-up) presented in tabular form.

# 5.8.1.1 Visit 1 (Screening, up to Day -28)

Prior to the initiation of study-specific screening assessments the Investigator or designee must provide the patient(s) a complete explanation of the purpose and evaluations (procedures and assessments) of the study. Subsequently, the patient must sign and receive a copy of an Informed Consent Form and authorization of use and disclosure of protected health information (PHI) that was approved by the institutional review board (IRB). Once informed consent has been obtained, the eligibility of the patient will be determined, and Screening Period assessments will be performed.


- Signed informed consent
- Complete medical history
- Physical examination
- Height and weight
- Concomitant medication assessment
- Vital signs (temperature, blood pressure, and pulse rate)
- Serum Pregnancy test (for women of childbearing potential)
- 12-lead ECG
- Clinical laboratory assessments including hematology, chemistries, and urine analysis

## 5.8.1.2 Visit 2- Day of Surgery (Day 1):

- Updated medical history and physical exam
- Concomitant medications assessment
- Clinical laboratory and vital sign assessments will be performed.
- Urine pregnancy test (for women of childbearing potential)
- 12- Lead ECG will be collected at least 15 minutes prior to infusion, and at least 15 minutes prior to surgery after infusion of OTL38 is completed
- A single dose of OTL38 will be infused IV over 60 minutes and will be completed at least one hour prior to initiation of intraoperative imaging and the time will be recorded
- AEs will be recorded during infusion of OTL38
- During and post-surgery any AEs and ADEs will be recorded.



#### Day 1 - Surgery

This is a phase 2, multi-center, single dose, open-label, exploratory study in suspected lung cancer patients scheduled to undergo endoscopic or thoracic surgery per CT/PET imaging based on standard of care.















# 5.8.1.3 *Visit 3-Follow-up (Day 7* $[\pm 4]$ ):

- Follow-up will be scheduled for Day 7 (± 4) on site
- AEs, ADEs, and concomitant medication information will be recorded.
- Clinical laboratory and vital sign assessments will be performed.

## 5.8.1.4 *Visits 4-Follow-up (Day 28 [\pm 4]):*

- Follow-up will be scheduled for Day 28 (±4) either via patient telephone interview or clinic visit
- AEs, ADEs, and concomitant medication information will be collected.


## 5.8.2 Surgical Reporting Schematic



## 5.8.3 Post-Surgery Questionnaire

After each surgery, the Investigator will fill out the questionnaire per Appendix 7.

# 5.8.4 Pathology Samples

All excised lesions will be processed as outlined in "Post-Surgery Tissue Processing". Please refer to the site manual for additional details.

## 5.8.5 Camera/Imaging System Exposure

A camera/imaging system will be used to identify tumor lesions under fluorescence prior to surgical excision of lesions, and again after surgical excision of lesions to identify persistent lesions. The Investigator will record the start and stop time for each exposure to fluorescence (pre-resection, post-initial resection, other [give reason]) in the eCRF only for in situ imaging. The total time of fluorescence will be calculated automatically.

| Status | Time On<br>Fluorescent Light | Time Off<br>Fluorescent Light |
|---|---|---|
| Before surgical excision | | |
| After initial surgical excision | | |
| Other (explain reason) | | |


#### 6 STUDY ENDPOINTS

# 6.1 Efficacy

The primary efficacy endpoints are the Sensitivity and False Positive rate of OTL38 for malignancy detection during Near Infrared Imaging (NIR).



# 6.2 Secondary Efficacy

The secondary efficacy endpoint is proportion of patients who demonstrate at least one CSE as a result of utilizing OTL-38 and Near Infrared Imaging.




# 6.3 Exploratory



# 6.4 Safety

- 1. Incidence rates of all treatment-emergent AEs (TEAEs) and ADEs from the time of OTL38 administration through follow-up Visit 4.
- 2. Laboratory parameters (chemistry and hematology) and vital signs collected at: screening, during day of surgery and 7-day follow-up
- 3. Electrocardiograms (ECG) and physical examinations will be collected at screening, day of surgery, and at least 24 hours after surgery.


#### 7 PROCEDURES FOR REPORTING ADVERSE EVENTS

#### 7.1 Adverse Events Definitions

The investigator will monitor the occurrence of AEs during the course of the study that will end with Visit 4.

The following definitions of terms are guided by the United States Code of Federal Regulations (21 CFR 312.32(a)) and are included here.

Adverse event is any untoward medical occurrence in a patient associated with the use of a drug in humans, whether or not considered drug related.

Suspected adverse reaction means any adverse event for which there is a reasonable possibility that the drug caused the adverse event. For the purposes of IND safety reporting, "reasonable possibility" means there is evidence to suggest a causal relationship between the drug and the adverse event. Suspected adverse reaction implies a lesser degree of certainty about causality than adverse reaction, which means any adverse event caused by a drug.

Unexpected adverse event (adverse drug experience) or (suspected) adverse reaction means any adverse event or (suspected) adverse reaction that is not listed in the investigator brochure or is not listed at the specificity or severity that has been observed.

An AE or suspected adverse reaction is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes: Death, a life- threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

An adverse event is considered "life-threatening" if, in the view of either the investigator or sponsor, its occurrence places the patient at immediate risk of death. It does not include an adverse event that, had it occurred in a more severe form, might have caused death.

Suspected Unexpected Serious Adverse Reaction (SUSAR) is any (suspected) adverse reaction (any adverse event for which there is a reasonable possibility that the drug caused the adverse event) that is both serious and unexpected.

#### 7.2 Adverse Device Effects Definitions

#### 7.2.1 Adverse Device Effect

An ADE is defined as any untoward and unintended response to a medical device, in this study, the camera/imaging system. This definition includes any event resulting from insufficiencies or inadequacies in the instructions for use or the deployment of the device, as well as any event that is the result of a user error [ISO 14155-1:2003 (E) 3.1].

All ADEs noted during the study will be reported in the eCRF.


## 7.2.1.1 Suspected Adverse Device Effect

A suspected ADE is a subset of all ADEs for which there is a reasonable possibility (i.e., evidence to suggest a causal relationship between the device and the ADE) that the device caused the event. Suspected ADE implies a lesser degree of certainty about causality than adverse device effect.

## 7.2.1.2 Unanticipated Adverse Device Effect

An unanticipated ADE is any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application, or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects [21 CFR 812.3 (s)].

# 7.3 Reporting of Adverse Events

#### 7.3.1 Adverse Events

The safety of all patients enrolled in this study will be recorded from the time of study drug administration and throughout the course of the study that will end with Visit 4.

All AEs will be recorded in the appropriate section of the eCRF. Patients withdrawn from the study because of AEs will be followed by the investigator until the outcome is determined. When appropriate, additional written reports and documentation will be provided.

All AEs beginning after the exposure to study drug must be reported to the sponsor or its designee if the onset of the AE was before Visit 4. All AEs that are judged by the investigator to be not related to study drug need not be reported to the sponsor or its designee after Visit 4. All AEs that are judged by the Investigator to be at least possibly related to study drug administration must be reported to the sponsor or its designee regardless of how much time has elapsed since the last exposure to study drug.

## 7.3.2 Laboratory Abnormalities

To the extent possible, all clinically significant laboratory abnormalities observed during the course of the study will be included under a reported AE describing a clinical syndrome (e.g., elevated blood urea nitrogen and creatinine in the setting of an AE of "renal failure" or elevated ALT/AST in the setting of an AE of "hepatitis"). In these cases (e.g., an AE of renal failure), the laboratory abnormality itself (e.g., elevated creatinine) does not need to be recorded as an AE.

In the absence of a reported AE identifying a clinical syndrome that encompasses the observed clinically significant laboratory abnormality that "isolated" laboratory abnormality itself should be reported as an AE.

Patients experiencing AEs or laboratory abnormalities will be assessed and appropriate evaluations performed until all parameters have returned to baseline levels, or are consistent with the patient's then-current physical condition, in the opinion of the investigator.


#### 7.3.3 Serious Adverse Events

Instructions for reporting Serious Adverse Events (SAE) and Suspected Unexpected Serious Adverse Reactions (SUSAR) are found on Page 2. A written report of all SAEs that occur after the administration of study drug and during the study (ending with Visit 4) must be submitted to the IRB/ethics committee (EC) and the Sponsor. SAEs/SUSARs must be reported to the Sponsor within 24 hours for a determination of expedited reporting to FDA, as described in Section 7.6. In all SAE reports, the investigator will advise whether or not the SAE is judged to be related to study drug administration. SAEs that occur after Visit 4 and are not reasonably associated with study drug do not require reporting per the instructions given below. All SAEs that are judged by the investigator to be at least possibly related to study drug administration must be reported to the sponsor or its designee regardless of how much time has elapsed since the last exposure to study drug. All AEs must be submitted to the IRB/EC in an annual report.

### 7.3.4 Reporting of Pregnancies

If a patient becomes pregnant during the course of the study, the investigator or site personnel must notify the Medical monitor (see Page 3 for details) within 5 working days after the investigator or site personnel become aware of the pregnancy. If an SAE occurs in conjunction with the pregnancy, then the reporting time frame for an SAE must be met.

# 7.3.5 Disease Progression

The progression of lung cancer (in patients diagnosed as such) per se will not constitute an AE. However, if the progression of the lung cancer meets the criteria for an SAE, then it should be reported as an SAE (see Page 2).

#### 1.1.1 Overdoses

Overdoses should be reported as a protocol violation. If an overdose results in an AE, the CRF AE page should be completed, and source documents included. If the overdose results in an SAE, then SAE reporting should be followed using the specific CRF pages with overdose information entered in the narrative section. All available clinical information relevant to overdose, including signs and symptoms, laboratory findings, and therapeutic measures or treatments administered, should be summarized and discussed.

# 7.4 Classification of Adverse Events by Severity

The investigator must categorize the severity of each AE according to the following:

- Mild: Awareness of signs or symptoms, but easily tolerated and are of minor irritant type.
   Symptoms do not require therapy or a medical evaluation; signs and symptoms are transient.
- Moderate: Events introduce a low level of inconvenience or concern to the participant, but are usually improved by simple therapeutic measures; moderate experiences may cause some interference with functioning


- Severe: Events generally require systemic drug therapy or other treatment; they are usually incapacitating
- Life-Threatening: Risk of imminent death requiring immediate intervention.

# 7.5 Classification of Adverse Events by Relationship to Study Drug Administration

The relationship of each AE to the study drug administration will be assessed by the investigator; after careful consideration, according to the following guidelines:

Definitely Related: An adverse event that has a timely relationship to the administration of the study drug and follows a known pattern of response for which no alternative cause is present

Probably Related: An adverse event that has a timely relationship to the administration of the study drug and follows a known pattern of response, but for which a potential alternative cause may be present

Possibly Related: An adverse event that has a timely relationship to the administration of the study drug, follows no known pattern of response, but a potential alternative cause does not exist

Not related: An adverse event for which there is evidence that it is definitely related to a cause other than the study; in general, no timely relationship to the administration of the drug exists, or if so, the event does not follow a pattern of response and an alternative cause is present

# 7.6 Adverse Events Qualifying for Expedited Reporting

All SUSARs, SAEs and unanticipated adverse device effects must be reported to On Target Laboratories or designee by telephone and in writing as soon as practical, but at least within 24 hours of initial report.

The investigator must report fatal and life-threatening SUSARs to the IRB within 7 calendar days of the initial receipt of information. On Target Laboratories or designee will report fatal and life-threatening SUSARs to the regulatory authorities and all investigators within 7 calendar days of the initial report of information.

The investigator must report non-fatal and non-life-threatening SUSARs to the IRB within 15 calendar days of the initial receipt of information. On Target Laboratories or designee will report non-fatal and non-life-threatening SUSARs to the regulatory authorities and all investigators within 15 calendar days of the initial report of information.

The investigator must report all unanticipated adverse device effects to the IRB within 10 calendar days of the initial receipt of information. On Target Laboratories or designee will report all unanticipated adverse device effects to the regulatory authorities and all investigators within 10 working days of the initial report of information.


# 8 DATA RECORDING, CRF PROCESSING, AND STATISTICAL ANALYSIS

# 8.1 Data Recording and CRF Processing

In place of recording patient data on paper CRFs, which will not be used in this study, site personnel are responsible for entering such data into the Electronic Data Capture (EDC) system. This system has been validated and is compliant with Food and Drug Administration (FDA), ICH, and European Union (EU) regulations and guidelines and with Department of Health and Human Services 21 CFR Part 11 rules for electronic records and electronic signatures.

#### 8.2 Statistical Methods

This is a phase 2, single dose, open-label exploratory study to estimate the safety and efficacy of OTL38 for intraoperative imaging of folate receptor positive lung nodules in patients diagnosed with FR+ adenocarcinoma of the lung, or with high clinical suspicion of lung nodule(s) warranting surgery based on CT and/or PET imaging. The primary objective of the study is to assess the safety of OTL38 in combination with fluorescent light imaging and to estimate the sensitivity and false positive rate.

Further analytic details for efficacy and safety will be provided in the statistical analysis plan (SAP).

## 8.2.1 Sample Size Estimation




## 8.2.2 Analysis Sets

The following definitions will be used to derive the analysis sets for the study.



**Safety Analysis Set (SAS):** The safety analysis set will include all patients exposed to OTL38 and/or the imaging system.

# 8.2.3 Description of Subgroups to be Analyzed

Using the FAS, descriptive summary statistics for the sensitivity, FPR, and CSE will also be provided for the following subgroups:

- Age: < 65 Yrs. Vs. ≥ 65 Yrs.
- Race/Ethnicity
- •
- Study Center




# 8.2.4 Patient Demographics, Baseline Disease Status, and Disposition

Descriptive statistics for patient demographics, baseline disease status, and patient disposition will be provided.

# 8.2.5 Statistical Analysis

# 8.2.5.1 Primary Efficacy Endpoints

The two co-primary efficacy endpoints are the sensitivity and false positive rate:






## 8.2.5.2 Secondary Efficacy Endpoint

The secondary efficacy endpoint is the proportion of patients with at efficacy endpoint,

## 8.2.5.3 Safety Evaluations

Safety will be evaluated using the safety analysis set and will include treatment emergent adverse events (TEAEs), adverse device effects (ADEs), serious adverse events (SAEs), vital signs, physical examinations, clinical laboratory measurements, electrocardiograms, and concomitant medications. For all safety assessments, the baseline value will be the last non-missing value recorded for a particular safety parameter before exposure to study drug. Treatment emergent adverse events are adverse events occurring during or after study drug exposure. Adverse device effects occur during or after exposure to the imaging device and classified as device effects by the Investigator. In general, the analysis of safety will be descriptive. No data will be imputed except for partial dates if required to determine if an adverse event is treatment emergent or a medication concomitant with exposure to study drug.

#### 8.2.5.3.1 Adverse Events and Adverse Device Effects

Adverse events occurring after the signing of informed consent but prior to exposure to OTL38 administration will be provided in line listings. Treatment emergent adverse events (TEAEs) will be summarized via the MedDRA system organ class and preferred term using subject incidence rates. Data will be tabulated by severity, physician assessment of the relationship to study drug, serious TEAEs, and TEAEs leading to death or study withdrawal. Further description of TEAEs may be defined by temporal onset to study drug infusion. Additional summaries of TEAEs identified as potential ADEs will also be provided.


#### 8.2.5.3.2 Clinical Laboratory Evaluations

The analysis of laboratory parameters will include descriptive statistics for the change from baseline to each post-baseline study visit as well as shifts from baseline to each post-baseline study visit for categorical lab parameters. In addition, shift tables (i.e., low-normal-high at baseline versus low-normal-high at last visit will be provided where appropriate. Urinalysis and pregnancy results will not be summarized but will be provided in a data listing. For all relevant laboratory data, values above or below normal limits will be flagged along with the direction of abnormality in line listings.

#### 8.2.5.3.3 *Vital Signs*

Vital signs will be summarized via descriptive statistics similar to that described above for clinical laboratory evaluations with regard to changes from baseline.

## 8.2.5.3.4 Physical Examination

Physical examination results will be provided in line listings only.

### 8.2.5.3.5 Electrocardiogram

Electrocardiogram results will be provided in line listings only.

#### 8.2.5.3.6 *Pathology and Immunohistochemistry*

Pathology and immunohistochemistry results will be provided in line listings.

## 8.2.5.4 Imaging System

Times on and off for the imaging system for each subject will be provided in line listings.

#### 8.2.5.5 Prior and Concomitant Medications

The prior and concomitant medications will be coded to identify the drug class and preferred drug name. Concomitant medications will include all medications that started, or were continuing, during or after administration of the study drug. Prior medications will include all recorded medications and supplements a patient was taking during the screening period that were stopped prior to administration of the study drug.

The number and percent of subjects using concomitant medications will be tabulated by drug class and preferred drug name for all subjects in the safety analysis set. If a subject has more than one medication within a drug class, the subject will be counted only once in that drug class. If a subject has more than one medication that codes to the same preferred drug name, the subject will be counted only once for that preferred drug name. All percentages will use the number of subjects in the safety analysis set as the denominator. The tabular summary will be sorted by descending order of overall incidence for concomitant medications only. Prior medications will be presented in line listings only. Concomitant medications will also be provided in line listings.


# 8.2.5.6 Handling of Missing Data, Subject Withdrawals, and Treatment Failures



In general, missing safety data will not be imputed with the possible exception of missing or partial dates. Details will be included in the SAP.

# 8.2.5.7 Interim Analyses

The data will be continuously monitored, but no formal interim analysis will be conducted.


### 9 ETHICS

The study will be conducted in compliance with applicable ICH guidelines, the ICH E6 GCP guideline, and regulations, guidelines, and applicable laws of the locale and countries where the study is conducted. The study will be conducted with the approval of a duly constituted IRB/EC in accordance with the requirement of United States regulation Title 21 CFR Part 56 - Institutional Review Boards. The nature and risks of the study will be fully explained to each patient and written consent obtained in accordance with the requirements of 21 CFR 50 - Protection of Human Subjects. Patients will be informed of their rights, including the right to withdraw from the study at any time.

# 9.1 Patient Information and Consent

A properly executed, written informed consent in compliance with national and local regulations and GCP guidelines will be obtained from each patient prior to entering the study or performing any study-related procedures that are not part of the patient's standard care. The Investigator will submit a copy of the informed consent document to the IRB/EC for review and approval before patients are enrolled. The Investigator will provide a copy of the signed informed consent to the patient and the original will be maintained in the patient's medical record.

#### 9.2 Institutional Review Board

The Investigator will provide the IRB/EC with all requisite material, including a copy of the protocol, IB, and the informed consent document. The study will not be initiated until the IRB/EC provides written approval of the protocol and the informed consent document and until approved documents have been obtained by the Investigator, and copies received by the Sponsor. Appropriate reports on the progress of this study by the Investigator will be made to the IRB/EC and the Sponsor in accordance with the applicable government regulations and in agreement with the Sponsor.


## 10 STUDY ADMINISTRATION

#### 10.1 Data

All information regarding the nature of the proposed investigation provided by the Sponsor or Study Monitor to the Investigator (with the exception of information required by law or regulations to be disclosed to the IRB, the patient, or the appropriate regulatory authority) must be kept in confidence by the Investigator.

All data recorded during the study must be available for audit against source data and for compliance with GCP and specific protocol requirements. Monitoring of the study progress and conduct will be ongoing. The Investigator will be responsible for the following:

- Monitoring study conduct to ensure that the rights of patients are protected;
- Monitoring study conduct to ensure trial compliance with GCP guidelines; and
- Monitoring accuracy, completion, and verification from source documents of study data.

## 10.2 Study Record Retention

US FDA regulations (21 CFR 312.62[c]) and the ICH Guideline for GCP (section 4.9 of that guideline) require that records and source documents pertaining to the conduct of this study and the distribution of investigational drug, including eCRFs, consent forms, laboratory test results, and medication inventory records, must be retained by the Investigator for 2 years after the last marketing application approval in an ICH region or for at least 2 years since formal discontinuation of clinical development of the investigational product. All state and local laws for retention of records also apply. The Investigator agrees to adhere to the document retention procedures by signing the protocol.

# 10.3 Patient Anonymity

The anonymity of participating patients must be maintained. Patients will be identified by their initials and an assigned patient number on CRFs, and other documents submitted to the Study Monitor. Documents that will not be submitted to the Study Monitor and that identify the patient (e.g., the signed informed consent document), must be maintained in strict confidence by the Investigator, except to the extent necessary to allow auditing by the appropriate regulatory authority, the Study Monitor, or Sponsor representatives.

#### 10.4 Publications

Following completion of the study, the results from the entire study, followed by the results from subsets of the study, may be reported at a scientific meeting and/or be published in a scientific journal. On Target Laboratories, Inc. will support these activities and will work with the Investigator(s) to determine how the meeting abstract, presentation and/or manuscript is written and edited, the number and order of authors, the meeting and/or journal to which it will be submitted, and other related activities. On Target Laboratories, Inc. acknowledges the right of the Investigator(s) to publish the results of this study after the entire study has been completed,


## 11 INVESTIGATOR'S STATEMENT

I have read the protocol entitled "A Phase 2, Single dose, Open-Label, Exploratory Study to Investigate the Safety and Efficacy of OTL38 Injection for Intraoperative Imaging of Folate Receptor Positive Lung Nodules" and agree that it contains all necessary details for carrying out the study as described. I will conduct this protocol as outlined therein and will make a reasonable effort to complete the study within the time designated. I will provide copies of the protocol and access to all information furnished by On Target Laboratories, Inc. to study personnel under my supervision. I will discuss this material with them to ensure they are fully informed about the drug and the study. I understand that the study may be terminated or enrollment suspended at any time by On Target Laboratories, Inc., with or without cause, or by me if it becomes necessary to protect the best interests of the study patients.

| Signature of Investigator | Date (day/month/year) |
|------------------------------|---------------------------------------|
| | · |
| Printed Name of Investigator | Site Number |


## 12 REFERENCES

Crane LMA, Arts HJG, van Oosten M, Low PS, van der Zee AGJ, van Dam GM, Bart J. The effect of chemotherapy on expression of folate receptor-alpha in ovarian cancer. Cell Oncol. 2012;35:9-18. doi: 10.1007/s13402-011-0052-6.

De Jesus EM, Keating JJ. Kularatne SA, Jiang JX, Judy R, Predina J, Nie S, Low P, Singhal S. Comparison of Folate Receptor Targeted Optical Contrast Agents for Intraoperative Molecular Imaging. International Journal of Molecular Imaging. 11 August 2015. PMID: 26491562. http://dx.doi.org/10.1155/2015/469047.

Keating JJ, Okusanya OT, DeJesus E, Judy RP, Jiang J, Deshpande C, Nie S, Low P, Singhal S. Intraoperative Molecular Imaging of Lung Adenocarcinoma Can Identify Residual Tumor Cells at Surgical Margins. Molecular Imaging and Biology. 2016 Apr;18(2):209-18. doi: 10.1007/s11307-015-0878-9. PMID: 26228697.

Leamon CP, Low PS. Membrane folate-binding proteins are responsible for folate protein conjugate endocytosis into cultured cells. Biochem J. 1993;291:855-60.

Okusanya OT, Deshpande C, Barbosa EM, Aggarwal C, Simone CB, Jiang J, Judy R, DeJesus E, Albelda S, Nie S, Low P, Singhal S. Molecular Imaging to Identify Tumor Recurrence Following Chemoradiation in a Hostile Surgical Environment. Molecular Imaging.

November 1, 2014;13:1-6.

Ross JF, Chaudhuri PK, Ratnam N. Differential regulation of folate receptor isoforms in normal and malignant tissues in vivo and in established cell lines. Physiologic and clinical implications. Cancer. 1994;73:2432–43.

SEER, US National Cancer Institute, Surveillance Epidemiology and End Results http://seer.cancer.gov/statfacts/html/ovary.html. Accessed 15 August 2014.

Shen J, Putt KS, Visscher DW, Murphy L, Cohen C, Singhal S, Sandusky G, Yang F, Dimitrov DS, Low PS. Assessment of Folate Receptor-β Expression in Human Neoplastic Tissues. Oncotarget. March 30, 2015;6(16):14700-9. doi: 10.18632/oncotarget.3739.

Stewart BW, Wild CP, editors. World Cancer Report 2014. Lyon, France: International Agency for Research on Cancer.

van Dam GM, Themelius G, Crane LMA, Pleijhuis RG, Kelder W, Sarantopoulos A, de Jong JS, Arts HJG, van der Zee AGJ, Bart J, Low PS, Ntziachristos V. Intraoperative tumor-specific fluorescence imaging in ovarian cancer by folate receptor-α targeting: first in-human results. Nature Med. 2011;17:1315-9.


# **APPENDICES**

| Appendix 1 | OTL38 Dose Preparation Manual | 55 |
|------------|-------------------------------|-----|
| Appendix 2 | Detailed Description of the | 58 |
| Appendix 3 | Detailed Description of the | 71 |
| Appendix 4 | Detailed Description of the | 82 |
| Appendix 5 | Detailed Description of the | 95 |
| Appendix 6 | Surgical Reporting Schematics | 107 |
| Appendix 7 | Investigator Questionnaire | 109 |


# Appendix 1 OTL38 Dose Preparation Manual







| <i>S</i> 5: | |
|-------------|----------------|
| | o- |
| | o <del>.</del> |


| <b>Appendix 2</b> Detailed Description of the |
|-----------------------------------------------|

















| a - |
|-----|






















| <br> |
|------|

**Appendix 3** Detailed Description of the














| 2 |
|---|
| - |

















| Appendix 4 Detailed Description of the |
|----------------------------------------|














| | 26 |
|-----|----|
| 100 | |

























| Appendix 5 | <b>Detailed Description of the</b> |
|------------|------------------------------------|














| <u> </u> |
|----------|








| -13 | |
|----------|----|
| <u> </u> | |
| | 1 |
| 32 | 25 |
| 32 | |


| - | |
|----|---|
| 32 | |
| | 8 |
| | * |


| × | V 16 |
|---|------|





Annendix 6 Surgical Reporting Schematics


## **Appendix 7** Investigator Questionnaire



